CLINICAL TRIAL: NCT06795464
Title: Effectiveness of Immersive Virtual Reality on Clinical Variables, Clinimetric Measurements, and Biomarkers in Patients with Persistent Shoulder Pain: a Randomized Multicenter Clinical Trial
Brief Title: Effectiveness of Immersive Virtual Reality on Biomarkers and Clinical and Clinimetric Variables in Patients with Persistent Shoulder Pain
Acronym: SHOULDERVR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Francisco de Vitoria (Other)
Responsible Party: Principal Investigator, Alberto Roldán, PhD, Universidad Francisco de Vitoria
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SHOULDERVIRTUALREALITY; UFV-2025/ (Other Grant/Funding Number: Universidad Francisco de Vitoria)
Record Dates: First submitted 2025-01-21; First posted 2025-01-28 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Shoulder Pain
Keywords: shoulder pain; virtual reality; exercise; randomized clinical trial; chronic pain
MeSH Terms: conditions — Shoulder Pain; Motor Activity; Chronic Pain | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (Active Comparator): Participants assigned to the control group will receive standard treatment for rotator cuff-related shoulder pain. This will consist of standardized therapeutic exercise performed for 25 minutes, 3 times per week, over a 12-week period. The exercise regimen will be individualized based on intensity, utilizing the Rate of Perceived Exertion (RPE) scale, with the goal of achieving intensity levels of 6-8 on a scale of 0 to 10
  Interventions: Procedure: Exercise
- Experimental group (Experimental): Participants in the experimental group will follow a treatment program that combines standard care with an immersive virtual reality (IVR) intervention. During the first 4 weeks, participants will undergo the IVR intervention, followed by the same standard treatment as the control group for the subsequent 8 weeks.
  IVR Intervention Protocol:
  Sessions and Equipment: Participants will attend up to 12 IVR sessions using a head-mounted device (HMD), the Meta Quest III, equipped with a hand-tracking system (Meta VR, Facebook, California) to enable interaction with the therapeutic software Dynamics PainRehab (Dynamics VR Rehab, Seville, Spain). The Meta Quest III HMD is chosen for its commercial availability, widespread use, minimal visual latency, and user-friendly interface. The software application, "Hombro PainRehab," features multisensory inputs (vision and sound), high-quality graphics, head and hand tracking, and provides a highly immersive experience. The IVR intervention incorporat
  Interventions: Device: Immersive Virtual Reality; Procedure: Exercise

INTERVENTIONS:
Device: Immersive Virtual Reality — Participants in the experimental group will follow a treatment program that combines standard care with an immersive virtual reality (IVR) intervention. During the first 4 weeks, participants will undergo the IVR intervention, followed by the same standard treatment as the control group for the subsequent 8 weeks.
  IVR Intervention Protocol:
  Sessions and Equipment: Participants will attend up to 12 IVR sessions using a head-mounted device (HMD), the Meta Quest III, equipped with a hand-tracking system (Meta VR, Facebook, California) to enable interaction with the therapeutic software Dynamics PainRehab (Dynamics VR Rehab, Seville, Spain). The Meta Quest III HMD is chosen for its commercial availability, widespread use, minimal visual latency, and user-friendly interface. The software application, "Hombro PainRehab," features multisensory inputs (vision and sound), high-quality graphics, head and hand tracking, and provides a highly immersive experience. The IVR intervention incorporate
  Other Names: virtual reality
  Arms: Experimental group
Procedure: Exercise — Participants assigned to the control group will receive standard treatment for rotator cuff-related shoulder pain. This will consist of standardized therapeutic exercise performed for 25 minutes, 3 times per week, over a 12-week period. The exercise regimen will be individualized based on intensity, utilizing the Rate of Perceived Exertion (RPE) scale, with the goal of achieving intensity levels of 6-8 on a scale of 0 to 10.

SUMMARY:
Shoulder pain is one of the primary reasons for seeking physiotherapy care. The high prevalence of rotator cuff-related shoulder pain underscores the need for research into novel treatment approaches that may enhance the clinical outcomes of conventional physiotherapy interventions.

Immersive Virtual Reality (IVR) has been demonstrated to serve as an effective adjunct for pain management by providing distraction and altering patients' pain perception. Specifically, when used alongside exercise, IVR has been shown to induce hypoalgesia in individuals with chronic low back pain. Additionally, IVR is emerging as a promising tool to enhance motivation and improve adherence to rehabilitation protocols, which is critical for long-term treatment implementation and achieving positive outcomes. These findings suggest that virtual reality may provide an innovative approach to managing pain in patients with rotator cuff-related shoulder pain, improving their pain experience, functionality, and quality of life.

To date, no study has directly compared the effectiveness of combining IVR with standard physiotherapy treatments versus standard treatments alone on clinical variables, clinimetric measures, and biomarkers in individuals with persistent shoulder pain related to the rotator cuff. Therefore, conducting a randomized multicenter clinical trial on this subject, facilitated by international collaboration among RIU-affiliated universities, could provide a robust foundation for implementing new technologies such as virtual reality in pain management and advancing rehabilitation strategies.

The objective of this project is as follows:

To compare the effectiveness of combining immersive virtual reality with standard physiotherapy treatment versus standard treatment alone on clinical variables, clinimetric measures, and biomarkers in individuals with persistent rotator cuff-related shoulder pain.

DETAILED DESCRIPTION:
Shoulder pain represents the third most common cause of musculoskeletal pain and the leading cause of non-traumatic upper limb pain. This condition holds significant musculoskeletal relevance, as up to 66.7% of individuals experience shoulder pain at least once in their lifetime, and symptoms persist beyond 18 months in 50% of cases, impacting daily activities at home and in the workplace. Furthermore, shoulder pain can disrupt sleep patterns and contribute to work-related challenges, such as sick leave, early retirement, or job loss. Persistent shoulder pain also imposes significant socioeconomic costs, estimated at $7 billion in the United States in 2000 and exceeding €1.5 million between 2004 and 2007 in the Canary Islands, Spain.

Physiotherapy has emerged as a promising approach for managing this condition. In Sweden, patients receiving physiotherapy as a first-line treatment generated lower total healthcare costs. Similarly, in the United States, musculoskeletal patients who initiated care with physiotherapy achieved better cost-effectiveness, required fewer sessions, and experienced greater functional recovery.

Diagnosing shoulder pain accurately remains challenging for clinicians, primarily due to inconsistencies and a lack of uniformity in diagnostic nomenclature and criteria. Consequently, diagnosis may need to rely on sub-classifications of patients with reliably reproducible characteristics. In this context, rotator cuff-related shoulder pain is consistently reported as the most prevalent diagnosis in individuals with shoulder pain.

Patients with rotator cuff-related shoulder pain often report moderate-to-severe pain intensity, limitations in daily activities, reduced range of motion, and/or loss of strength. Persistent pain in this condition is also commonly associated with psychosocial factors, such as fear of movement, pain hypervigilance, and/or loss of self-efficacy-barriers that can hinder recovery. Collectively, these factors significantly affect patients' quality of life.

A novel aspect of this project is the proposed examination of biomarkers associated with systemic inflammation and chronic pain in this clinical population, specifically C-reactive protein (CRP) and calcitonin gene-related peptide (CGRP). C-reactive protein is a marker of systemic inflammation, with elevated levels linked to various chronic pain conditions, suggesting an inflammatory component that may modulate pain perception and intensity in these patients. Meanwhile, CGRP is a neuropeptide involved in nociceptive signal transmission and inflammatory response modulation. Elevated CGRP levels have been documented in several chronic pain conditions, including osteoarthritis, migraines, and joint disorders, where peripheral and central sensitization processes are present.

In animal studies, CGRP has been shown to play a role in triggering neurogenic inflammation and its association with pain pathways. In conditions like rotator cuff-related shoulder pain, characterized by persistent pain, complex interactions between inflammatory processes and neurobiological mechanisms are likely to occur. Evaluating these biomarkers is particularly relevant to deepen our understanding of the underlying pathophysiological mechanisms in this patient population.

The use of virtual reality (VR) has emerged as an innovative strategy for managing patients with pain, disability, and reduced quality of life. On one hand, it can modulate the context of motor relearning, an aspect of particular relevance for individuals with persistent shoulder pain, where strength and mobility deficits are common. On the other hand, the hypoalgesic mechanisms underlying the effects of VR are multifactorial, mediated by various dimensions of the pain experience, including sensory-discriminative, affective-motivational, and evaluative-cognitive aspects, as well as motor behavior itself.

Moreover, VR appears to modulate pain perception by stimulating auditory, visual, and sensorimotor neural networks and activating descending inhibitory systems, thereby influencing pain perception. Interestingly, severe pain and disability, rather than being contraindications, may serve as indications for implementing VR.

This therapeutic approach can also be tailored to the individual needs of patients, considering factors such as functional levels, social context, and age, which may influence adaptability to the technology and, consequently, treatment adherence and outcomes.

Finally, VR has demonstrated its potential as a high-quality, cost-effective treatment option for chronic low back pain, highlighting its capacity to provide an accessible and effective alternative that reduces the economic burden on healthcare systems and patients alike.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 70 years.
* Shoulder pain persisting for at least six months.
* Presence of shoulder pain during movement.
* Clinical diagnosis of rotator cuff-related shoulder pain.
* Willingness to participate in the study and signing of informed consent.

Exclusion Criteria

* Shoulder pain related to cervical spine conditions.
* Presence of pain in the elbow, wrist, and/or hand.
* Clinical diagnosis of frozen shoulder.
* Clinical diagnosis of shoulder instability.
* Cognitive impairments.
* Concomitant physiotherapy treatments during the study period.
* History of trauma associated with the onset of shoulder pain.
* Previous fractures in the affected shoulder.
* Prior surgeries in the affected shoulder.
* Use of analgesic or anti-inflammatory medications within 24 hours prior to study participation.

Presence of rheumatic or neurological diseases.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-12-20 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Pain | Baseline, 1, 2 and 3 months follow-up
  Pain intensity will be assessed using the Numeric Pain Rating Scale (NPRS), a visual 11-point scale ranging from 0 (no pain) to 10 (worst imaginable pain).
Shoulder disability | Baseline, 1, 2 and 3 months follow-up
  Self-reported shoulder function will be evaluated using the Spanish version of the Shoulder Pain And Disability Index (SPADI). This questionnaire, originally developed to assess shoulder pain and disability through 13 items (Williams et al., 1995), has been described as a tool capable of effectively discriminating between patients with improving or worsening conditions (Roy et al., 2009). Following a transcultural adaptation, the Spanish version (Membrilla-Mesa et al., 2015) retains the 13 items, assessing pain and disability in shoulder dysfunction. This patient-reported outcome measure is suitable for both clinical practice and research.
Shoulder external rotation strength | Baseline, 1, 2 and 3 months follow-up
  Isometric shoulder strength in external rotation will be measured using a MicroFET 2 MT Digital Handheld Dynamometer (Hoggan Health Industries, West Draper, UT). Handheld dynamometry has demonstrated good-to-excellent intra-examiner reliability for measuring isometric shoulder strength (Intraclass Correlation Coefficient = 0.87-0.99) (McLaine et al., 2016; Holt et al., 2016).
Handgrip strength | Baseline, 1, 2 and 3 months follow-up
  Handgrip strength will be assessed using a Jamar Hand Dynamometer (Sammons Preston Rolyan, Bolingbrook, IL). This device has shown good-to-excellent intra-examiner reliability for measuring isometric handgrip strength (Intraclass Correlation Coefficient = 0.85-0.98) (Roberts et al., 2011).
Shoulder mobility | Baseline, 1, 2 and 3 months follow-up
  Shoulder mobility will be assessed during movements of flexion, abduction, external rotation at 0° abduction, external rotation at 90° abduction, and internal rotation at 90° abduction. Measurements will be conducted using a smartphone application-based inclinometer (Plaincode Software Solutions, Gunzenhausen, Germany), which has been validated with excellent inter-examiner reliability and validity in symptomatic individuals (Intraclass Correlation Coefficient > 0.80) (Werner et al., 2014).

SECONDARY OUTCOMES:
Biomarkers | Baseline, 1 and 3 months follow-up
  A blood sample will be collected from the antecubital vein, which will subsequently undergo centrifugation, aliquoting, and storage at -80°C until analysis. This procedure will be conducted in the Exercise Physiology Research Laboratory of UFV by nurses from the external laboratory Eurofins Megalab, who will be responsible for the collection and analysis of biological samples.
  The blood markers to be evaluated in the participants include:
  Oxidative stress and inflammation biomarkers: C-reactive protein (CRP). Neurobiological markers associated with chronic pain processes: calcitonin gene-related peptide (CGRP).
Quality of life | Baseline, 1, 2 and 3 months follow-up
  Quality of life will be assessed using the SF-12 (Short Form Health Survey), which evaluates eight health dimensions related to perceived quality of life. The SF-12 has been shown to be a reliable and valid instrument in diverse populations (Ware et al., 1996).
Kinesiophobia | Baseline, 1, 2 and 3 months follow-up
  Fear of movement will be measured using the Tampa Scale for Kinesiophobia (TSK). This scale evaluates fear of movement and has demonstrated high reliability and internal consistency (Intraclass Correlation Coefficient = 0.76-0.90) (Vlaeyen et al., 1995).
Daily Activity Avoidance Behaviors | Baseline, 1, 2 and 3 months follow-up
  Daily activity avoidance behaviors will be assessed with the Shoulder Activity Daily Avoidance Photographic Scale (Shoulder ADAP Scale) (Ansanello et al., 2022). This scale includes 15 photographs distributed across three domains, assessing pain-related activity avoidance in individuals with unilateral or bilateral shoulder pain. Scores range from 0 to 100 (0 = no avoidance, 100 = extreme avoidance), with 15 items distributed as follows:
  Free Movement (5 items): Total = [(sum × 10)/5] High Effort (7 items): Total = [(sum × 10)/7] Self-Care (3 items): Total = [(sum × 10)/3] The total score is calculated as Total = [(sum × 10)/15]. The Shoulder ADAP Scale has shown internal consistency values of 0.92 for free movement (factor 1), 0.89 for high effort (factor 2), and 0.92 for self-care (factor 3), with excellent test-retest reliability (ICC = 0.94) across all domains and the total score (Ansanello et al., 2023; Scaglione et al., 2024).
Pain hypervigilance | Baseline, 1, 2 and 3 months follow-up
  Pain hypervigilance will be assessed using the Pain Vigilance and Awareness Questionnaire (PVAQ), a tool designed to measure attention and vigilance to pain. The PVAQ has demonstrated high internal reliability and validity in various clinical contexts (McCracken, 1997).
Self efficacy | Baseline, 1, 2 and 3 months follow-up
  Self-efficacy will be measured using the Pain Self-Efficacy Questionnaire (PSEQ), which evaluates patients' confidence in their ability to perform activities despite pain. The PSEQ has shown excellent reliability and validity in populations with chronic pain (Nicholas, 2007).
Motor and functional deficits related to pain | Baseline, 1, 2 and 3 months follow-up
  Motor and functional deficits related to pain will be assessed using the 16-item version of the Biobehavioral Pain and Movement Questionnaire (CBioD-MOV). This tool evaluates four major subscales: physical activity self-efficacy, disability, movement avoidance behavior, and perceived functional capacity. The CBioD-MOV uses a 5-point Likert scale and scores range from 0 to 62. The psychometric adaptation of the Spanish version has shown good-to-excellent reliability for Standard Error of Measurement (SEM) and Minimal Detectable Change (MDC) (La Touche et al., 2024).
Implicit motor imagery performance | Baseline, 1, 2 and 3 months follow-up
  Implicit motor imagery performance will be evaluated using a left/right judgment task. Participants will view a series of shoulder images displayed on a computer screen and determine whether the images depict a left or right shoulder. This test has shown adequate reliability (Breckenridge et al., 2017). The task will be performed using the Recognise™ software (noigroup.com, Adelaide, Australia), where participants will complete a block of 30 randomized images of shoulders in various postures and rotations. Participants must identify the correct side as quickly and accurately as possible by pressing the corresponding key on the screen.
Sleep quality | Baseline, 1, 2 and 3 months follow-up
  Sleep quality will be estimated using the Oviedo Sleep Questionnaire (COS), designed to assess sleep disorders, particularly insomnia and hypersomnia. The COS consists of 15 items, 13 of which are grouped into three subscales:
  Subjective Sleep Satisfaction: Item 1 (scored 1-7). Insomnia: Items 2-1, 2-2, 2-3, 2-4, 3, 4, 5, 6, 7 (scored 1-5; total range: 9-45).
  Hypersomnia: Items 2-5, 8, 9 (scored 1-5). Two additional items provide information on the use of sleep aids and adverse sleep events. Higher scores in the insomnia subscale indicate greater severity. The COS has demonstrated adequate concurrent validity and reliability (Bobes et al., 1998).

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Francisco de Vitoria, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided
At this time, there are no plans to share individual participant data (IPD). The primary reason for this decision is to protect the confidentiality and privacy of participants, as sharing IPD may pose a risk of re-identification despite anonymization efforts. Additionally, the study does not have a specific framework or infrastructure in place for secure and compliant IPD sharing.
  However, summary data and results of the study will be disseminated through peer-reviewed publications and presentations at scientific conferences, ensuring that the scientific community and the public can benefit from the findings.

REFERENCES:
- [Background] Ahmadpour N, Randall H, Choksi H, Gao A, Vaughan C, Poronnik P. Virtual Reality interventions for acute and chronic pain management. Int J Biochem Cell Biol. 2019 Sep;114:105568. doi: 10.1016/j.biocel.2019.105568. Epub 2019 Jul 12. PMID 31306747